CLINICAL TRIAL: NCT02071680
Title: Cardiac Mapping of Autonomic Atrial Innervation and Its Relation to MIBG Nuclear Imaging in Patients With Atrial Fibrillation
Brief Title: Autonomic Innervation and MIBG Imaging
Acronym: MIBG-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Robert Lemery, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140815-01H
Record Dates: First submitted 2014-01-15; First posted 2014-02-26 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial cardiac innervation; catheter ablation of atrial fibrillation; High Frequency Stimulation; ganglionated plexuses; 123I-mIBG; nuclear imaging
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iodine-123 Meta-iodobenzylguanidine (Other): 123I-mIBG administration followed by nuclear imaging pre-ablation and post-ablation
  Interventions: Other: Iodine-123 Meta-iodobenzylguanidine

INTERVENTIONS:
Other: Iodine-123 Meta-iodobenzylguanidine — A single injection of the 123I-mIBG will be given. Imaging will be done twice following injection: at 0120 minutes and 3-5 hours. The timing is dependent on the specific participant and imaging characteristics.
  The imaging is done for approximately 24 minutes at each time point.
  Other Names: 123I-mIBG

SUMMARY:
Patients with symptomatic atrial fibrillation (AF), a rapid beating of the upper heart chambers, can undergo catheter ablation to control or eliminate their rhythm disorder. The radiopharmceutical 123I-mIBG (Adreview™ GE Healthcare) has been introduced to visually identify cardiac innervation. This study will use non-invasive evaluation using MIBG imaging to study if we can predict baseline autonomic characteristics in patients with AF, as well as clinical outcome based on post ablation imaging

DETAILED DESCRIPTION:
This is a single centre, interventional, Phase III trial using the radiopharmaceutical 123I-mIBG for imaging. In this pilot study, up to 7 eligible participants will undergo pre-ablation and post ablation nuclear imaging.

The major objective of our study is to evaluate the relationship between non-invasive imaging of cardiac innervation with invasive mapping of atrial innervation as determined by High Frequency Stimulation (standard of care to physiologically document autonomic function). This will be followed by the clinical ablation procedure, as discussed by the cardiac electrophysiologist, consisting of pulmonary vein (PV) antral isolation, inclusive of regions of autonomic innervation, and sites showing complex fractionated atrial electrograms (CFAE) when clinically indicated.

The secondary objective is to determine the relationship between catheter ablation of AF and non-invasive nuclear imaging of cardiac innervation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Symptoms including one or more of the following: palpitations, shortness of breath, dizziness, presyncope or syncope, chest pain, tiredness or lack of energy.
* Failure of beta-blockers or at least one antiarrhythmic agent other than Amiodarone to prevent AF. In those patients who are not eligible to antiarrhythmic agents other than Amiodarone, patients may choose to undergo catheter ablation rather than starting Amiodarone.
* Paroxysmal (self-terminating AF within 7 days) or persistent AF (requiring an intervention to terminate or lasting more than 7 days).

Exclusion Criteria:

* Intracardiac thrombus as determined by transesophageal echocardiography
* Class III or IV congestive heart failure
* Persistent AF duration of more than 3 years
* Myocardial infarction within the last 6 months
* Left atrial size of greater than 55 mm determined by 2D echocardiogram
* Inability to undergo a transesophageal echocardiogram or cardiac CT
* Inability to undergo D-SPECT™ imaging
* Inability to take Warfarin or the new oral anticoagulants
* Previously received 123I-mIBG or 131I-mIBG
* History or suspicion of significant allergic reaction or anaphylaxis to iodine or iodinated imaging agents
* Use of medications for non-cardiac medical conditions that are known to interfere with 123I-mIBG uptake and these medications cannot be safely withheld for at least 24 hours before study procedures
* Diagnosis of or signs or symptoms of a neurologic disease such as Parkinson's disease, multiple systems atrophy or Parkinsonian syndromes, or other diseases known to affect the sympathetic nervous system
* Pregnancy as determined by a pre-procedure pregnancy tests

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Concordance | 2 years
  The concordance of the 123I-mIBG visual images with the identification of autonomic sites as determined by high frequency stimulation (HFS).

SECONDARY OUTCOMES:
Observation of effects | 2 years
  The effects of radiofrequency ablation of AF on cardiac innervation will be observed visually on 123l-mlBG images and clinically with participant follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lemery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Lemery R, Birnie D, Tang AS, Green M, Gollob M. Feasibility study of endocardial mapping of ganglionated plexuses during catheter ablation of atrial fibrillation. Heart Rhythm. 2006 Apr;3(4):387-96. doi: 10.1016/j.hrthm.2006.01.009. Epub 2006 Feb 28. PMID 16567283
- [Background] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504
- Available data/document: Published article — http://www.heartrhythmjournal.com/article/S1547-5271(16)30735-4/fulltext — DOI: http://dx.doi.org/10.1016/j.hrthm.2016.08.038